CLINICAL TRIAL: NCT04911868
Title: Surgical Management During the Era of COVID-19 at a Private Tertiary Care Hospital of Karachi, Pakistan: A Cross Sectional Study
Brief Title: Surgical Management During the Era of COVID-19
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Ather Enam, Professor, Aga Khan University
Other Study IDs: 2020-5014-11563.
Record Dates: First submitted 2021-05-31; First posted 2021-06-03 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: COVID 19
Keywords: COVID 19; Pandemic,; Surgery,; Management,; Guidelines
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Lower middle-income countries (LMICs) like Pakistan with limited health care facilities the gravity of COVID 19 is severe. Effective management and implementation of processes and planning is imperative. In surgical procedures additional time is required to prepare for surgery in a suspected/confirmed case of COVID-19 in daily routines regardless of whether surgery would happen. Therefore, for effective management of surgical procedures the Aga Khan University, Karachi, Pakistan has established a COVID testing algorithm for effective management of the surgical patients.

The objectives of the study are

1. To evaluate the outcomes of COVID testing algorithm established for surgery patients presenting to Aga Khan University Karachi, Pakistan
2. To compare the outcomes among patients who underwent elective versus emergency surgery.

DETAILED DESCRIPTION:
The disease declared as corona virus disease 2019 (COVID-19) by the World Health Organization was initially known as severe acute respiratory syndrome corona virus 2 (SARS-CoV-2). It is caused by a single-stranded RNA virus that belongs to the corona virus family known as 2019-nCoV (SARS-CoV-2). The disease is highly contagious and transmitted mainly by droplets or close contact. The first case occurred in Wuhan, Hubei Province, China in December 2019 . On March 11, 2020, WHO declared COVID-19 as a pandemic disease and by March 26, 2020, it had spread to almost 199 countries and territories worldwide with more than 462680 cases and around 20834 deaths . The COVID-19 pandemic reached Pakistan on 26 February 2020, when a student in Karachi tested positive upon returning from Iran. By 18 March, cases had been registered in all four provinces. With a total of 3277; in Punjab there were 1493 cases, Sindh (881), Khyber Pakhtunkhwa (405) and Balochistan (191), Gilgit Baltistan (210), Azad Jammu and Kashmir (15) and Federal (ICT) (82).

As the global incidence of COVID-19 disease is increasing in different parts of the world the COVID-19 pandemic has disrupted the health care services , in terms of its capability to manage affected people and the ability to provide standard treatment for critically ill patients in a safe environment . Similarly, the surgical procedures are minimized or temporarily suspended to address the overwhelming and devastating increase in COVID-19 patient care needs. However, decisions regarding surgical intervention in this resource scarce time must undergo rigorous ethical and clinical evaluation . In this era, it is essential that all the health care providers must execute standardized essential perioperative measures including the use of Personal Protective Equipment (PPEs) to control disease transmission and avoid unwanted complications. All patients need to be managed as COVID-19 patients till confirmed by results. Elective procedures are recommended to be postponed and to consider only urgent, lifesaving procedures and oncologic surgeries that are associated with worse outcome if delayed.

In a Lower middle-income countries (LMICs) like Pakistan with limited health care facilities the gravity of COVID 19 is severe. Effective management and implementation of processes and planning is imperative. In surgical procedures additional time is required to prepare for surgery in a suspected/confirmed case of COVID-19 in daily routines regardless of whether surgery would happen. Therefore, for effective management of surgical procedures the Aga Khan University, Karachi, Pakistan has established a COVID testing algorithm for effective management of the surgical patients.

It was a cross sectional study conducted at the Aga Khan University Hospital Karachi, Pakistan, Department of Surgery. Nonprobability consecutive sampling technique was employed to recruit patients . The data for the study was collected on a Proforma from the patients' medical records from May 2020 onwards. The data was collected on patients' demographic, type of case (elective, orange or red), type of surgery, COVID screening (non-suspected or suspected case), COVID results (positive negative) and surgery outcome, classification of surgery according to specialties.

Ethical exemption was sorted. All the patient information was kept in lock and key. The data base was password protected and was only accessible by the research team. All the patient information was deidentified. When the patients were admitted to the hospital consent was taken from them, they were informed that their information will be used for research purpose and the study results will be published in group form and no individual information will be disclosed The data was analyzed by using SPSS version 22. Descriptive for qualitative variables was reported as frequency and percentages and was assessed by chi-square and fisher exact test. Bars charts for categorical variables and histogram/ line graphs were presented for quantitative variables. A p value of <0.05 was kept significant throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for surgical procedures to Aga Khan University Hospital from May 2020 onwards were included

Exclusion Criteria:

* Patients who left against medical advice (LAMA)
* Patients with missing information

Ages: 1 Year to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting for surgical procedures to Aga Khan University Hospital from May 2020 onwards were included
Sampling Method: Non-Probability Sample
Enrollment: 6846 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
The patients who underwent elective versus emergency surgery. 2. Frequency of Covid positive patients who underwent surgery or the surgery was deferred. the outcomes among patients who underwent elective versus emergency surgery. | May to October 2020
Frequency of Covid positive and negative patients presenting for surgery | May to October 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Al-Balas M, Al-Balas HI, Al-Balas H. Surgery during the COVID-19 pandemic: A comprehensive overview and perioperative care. Am J Surg. 2020 Jun;219(6):903-906. doi: 10.1016/j.amjsurg.2020.04.018. Epub 2020 Apr 18. No abstract available. PMID 32334800
- [Background] Zacharia BE, Eichberg DG, Ivan ME, Hanft S, Boockvar JA, Isildak H, Mansouri A, Komotar RJ, D'Amico RS. Letter: Surgical Management of Brain Tumor Patients in the COVID-19 Era. Neurosurgery. 2020 Aug 1;87(2):E197-E200. doi: 10.1093/neuros/nyaa162. No abstract available. PMID 32347942
- [Background] Proietti S, Gaboardi F, Giusti G. Endourological Stone Management in the Era of the COVID-19. Eur Urol. 2020 Aug;78(2):131-133. doi: 10.1016/j.eururo.2020.03.042. Epub 2020 Apr 14. No abstract available. PMID 32303384